CLINICAL TRIAL: NCT01032109
Title: Verteporfin Photodynamic Therapy Alone Versus Combined With Intravitreal Bevacizumab for Neovascular Age-related Macular Degeneration
Brief Title: Photodynamic Therapy Alone Versus Combined With Intravitreal Bevacizumab for Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Takahiro Kawaji, Associate Professor, Kumamoto University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCBK610
Record Dates: First submitted 2009-12-12; First posted 2009-12-15 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — A single intravitreal injection of 1.25 mg of bevacizumab (0.05 mL of solution prepared from Avastin, 100 mg/4 mL vial) was performed within 2 weeks after PDT treatment.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to compare 12-month results of two single initial treatments-photodynamic therapy with verteporfin alone and this therapy combined with intravitreal bevacizumab-for neovascular age-related macular degeneration, not including patients with polypoidal choroidal vasculopathy who were presumed to have age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* choroidal neovascularization caused by age-related macula degeneration
* no previous treatment
* a follow-up at least 12 months
* a baseline visual acuity ranging from a letter score of 0 to 70 on the Early Treatment Diabetic Retinopathy Study chart

Exclusion Criteria:

* choroidal neovascularization caused by other eye diseases
* ocular surgery within the past 3 mouths
* history of uveitis
* intraocular pressure higher than 25 mmHg, or glaucoma
* history of systemic or ocular thromboembolic events.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Visual acuity | The comparison between baseline and 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kawaji, MD, PhD, Principal Investigator — Department of Ophthalmology, Kumamoto University Graduate School & Medical Sciences
Locations (1):
- Department of Ophthalmology and Visual Science, Graduate School of Medical Sciences, Kumamoto University, Kumamoto, Japan

REFERENCES:
- [Derived] Hara R, Kawaji T, Inomata Y, Tahara J, Sagara N, Fukushima M, Tanihara H. Photodynamic therapy alone versus combined with intravitreal bevacizumab for neovascular age-related macular degeneration without polypoidal choroidal vasculopathy in Japanese patients. Graefes Arch Clin Exp Ophthalmol. 2010 Jul;248(7):931-6. doi: 10.1007/s00417-010-1343-8. Epub 2010 Mar 10. PMID 20221623